CLINICAL TRIAL: NCT01832688
Title: Assessment of the Nutritional Status of Pregnant Women in Zinder, Niger and Optimization of Prenatal Care Services
Brief Title: Assessment of the Nutritional Status of Pregnant Women and Optimization of Prenatal Care Services
Status: Completed | Type: Observational
Sponsor: University of California, Davis (Other)
Collaborators: Helen Keller International (Other); Micronutrient Initiative (Other)
Responsible Party: Sponsor
Other Study IDs: 447971; 10-1335-UCALIF (Other Grant/Funding Number: The Micronutrient Initiative)
Record Dates: First submitted 2013-04-04; First posted 2013-04-16 (Estimated); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Pregnancy
Keywords: iron and folic acid supplements; anemia; gestational weight gain
MeSH Terms: conditions — Anemia; Gestational Weight Gain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and urine sample for assessment of nutritional status
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Baseline cohort: The baseline survey will be implemented among pregnant women in randomly selected villages using a continuous enrollment schedule over the period of 18 months
- Optimization cohort: The programmatic impact of optimized prenatal care services on women's health and behavior will be assessed among pregnant women in randomly selected villages (Programmatic prenatal care optimization)
  Interventions: Other: Programmatic prenatal care optimization

INTERVENTIONS:
Other: Programmatic prenatal care optimization — To further integrate and improve nutrition-related services and messages in the prenatal care package.
  Groups: Optimization cohort

SUMMARY:
A national survey in Niger found that women and children are at risk of undernutrition and that many pregnant women don't visit health centers during pregnancy as often as is recommended. The aim is to assess the nutritional and health status of pregnant women in the Zinder region and to understand their knowledge, attitudes and practices related to health and nutrition during pregnancy. In collaboration with the Medical District of Zinder the prenatal care services will be optimized and the programmatic impact on gestational weight gain and anemia prevalence will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant

Exclusion Criteria:

* Pregnant women, who have severe illness warranting immediate hospital referral

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women residing in participating villages
Sampling Method: Non-Probability Sample
Enrollment: 2306 (Actual)
Dates: Start 2014-02; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Prevalence of inadequate gestational weight gain | 6 months
Anemia prevalence | 6 months
Access and adherence to prenatal iron and folic acid supplements | 6 months

SECONDARY OUTCOMES:
Prevalence of inadequate dietary diversity scores | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sonja Y Hess, PhD, Principal Investigator — University of California, Davis
Locations (1):
- Helen Keller International, Zinder, Niger

REFERENCES:
- [Background] Hess SY, Ouedraogo CT, Bamba IF, Wessells KR, Keith N, Faye T, Ndiaye B, Doudou M, Nielsen J. Using formative research to promote antenatal care attendance and iron folic acid supplementation in Zinder, Niger. Matern Child Nutr. 2018 Apr;14(2):e12525. doi: 10.1111/mcn.12525. Epub 2017 Sep 19. PMID 28924978
- [Background] Wessells KR, Young RR, Ferguson EL, Ouedraogo CT, Faye MT, Hess SY. Assessment of Dietary Intake and Nutrient Gaps, and Development of Food-Based Recommendations, among Pregnant and Lactating Women in Zinder, Niger: An Optifood Linear Programming Analysis. Nutrients. 2019 Jan 2;11(1):72. doi: 10.3390/nu11010072. PMID 30609695
- [Result] Wessells KR, Ouedraogo CT, Young RR, Faye MT, Brito A, Hess SY. Micronutrient Status among Pregnant Women in Zinder, Niger and Risk Factors Associated with Deficiency. Nutrients. 2017 Apr 26;9(5):430. doi: 10.3390/nu9050430. PMID 28445440
- [Result] Begum K, Ouedraogo CT, Wessells KR, Young RR, Faye MT, Wuehler SE, Hess SY. Prevalence of and factors associated with antenatal care seeking and adherence to recommended iron-folic acid supplementation among pregnant women in Zinder, Niger. Matern Child Nutr. 2018 Feb;14 Suppl 1(Suppl 1):e12466. doi: 10.1111/mcn.12466. PMID 29493896
- [Result] Hess SY, Ouedraogo CT, Young RR, Bamba IF, Stinca S, Zimmermann MB, Wessells KR. Urinary iodine concentration identifies pregnant women as iodine deficient yet school-aged children as iodine sufficient in rural Niger. Public Health Nutr. 2017 May;20(7):1154-1161. doi: 10.1017/S1368980016003232. Epub 2016 Dec 15. PMID 27974077
- [Result] Ouedraogo CT, Wessells KR, Young RR, Bamba IF, Faye MT, Banda N, Hess SY. The mixed effects of a package of multilevel interventions on the health and care of pregnant women in Zinder, Niger. BMJ Glob Health. 2019 Dec 10;4(6):e001200. doi: 10.1136/bmjgh-2018-001200. eCollection 2019. PMID 31908852
- [Result] Ouedraogo CT, Wessells KR, Young RR, Faye MT, Hess SY. Prevalence and determinants of gestational weight gain among pregnant women in Niger. Matern Child Nutr. 2020 Jan;16(1):e12887. doi: 10.1111/mcn.12887. Epub 2019 Sep 30. PMID 31568674
- [Derived] Ouedraogo CT, Vosti SA, Wessells KR, Arnold CD, Faye MT, Hess SY. Out-of-pocket costs and time spent attending antenatal care services: a case study of pregnant women in selected rural communities in Zinder, Niger. BMC Health Serv Res. 2021 Jan 8;21(1):47. doi: 10.1186/s12913-020-06027-2. PMID 33419448